CLINICAL TRIAL: NCT03269227
Title: Accelerated Hypofractionated Radiotherapy in the Treatment of Malignant Pleural Mesothelioma
Acronym: MesoRT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRST163.01
Record Dates: First submitted 2017-08-16; First posted 2017-08-31 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: Malignant Pleural Mesothelioma; Radiotherapy; Tomotherapy; Hypofractionation
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Accelerated hypofractionation with Tomotherapy (Experimental): Tomotherapy Treatment Planning System (TPS) will be used for treatment plannings.
  Patient' set-up daily control through Tomo-image (CT megavoltage) immediately before each sitting of all the patients.
  Prescription dose to the target: 30 Gy in 5 daily fraction (at the reference isodose 60-70%) with an internal increasing inhomogenous dose of up to 37.5 Gy-40 Gy for Gross Tumor Volume (GTV).
  Interventions: Radiation: Accelerated hypofractionation with Tomotherapy

INTERVENTIONS:
Radiation: Accelerated hypofractionation with Tomotherapy — Tomotherapy TPS will be used for treatment plannings. Patient' set-up daily control through Tomo-image (CT megavoltage) immediately before each sitting of all the patients.
  Prescription doses:
  Prescription dose to the target: 30 Gy in 5 daily fraction (at the reference isodose 60-70%) with an internal increasing inhomogenous dose of up to 37.5 Gy-40 Gy for GTV.
  Steroids (methylprednisolone 4 mg daily) should be used from day 1 of radiotherapy to day + 30 after the end of the treatment.

SUMMARY:
This is a monocentric prospective study of radiotherapy using accelerated hypofractionation with Tomotherapy in Malignant Pleural Mesothelioma (MPM) patients after pleurectomy / decortication (P / D) or biopsy.

The treatment will be delivered using Tomotherapy, that allows to adopt dose accelerated hypofraction criteria. Treatment duration is 5 consecutive days.

DETAILED DESCRIPTION:
The role of radiation therapy remains to be defined in unresected MPM or after P/D. For the latter, local control remains the primary objective but radiotherapy (RT) is a challenge because of the risk of pneumonia in the intact lung. There are no specific clinical data to support the use of adjuvant radiation therapy after P/D or definitive radiation therapy after biopsy-based diagnosis for patients not amenable to surgery.

However, recent publications on Intensity Modulated Radiotherapy (IMRT) and conventional fractionation after P/D or biopsy have shown the feasibility and acceptable toxicity profile of the treatment.

The investigators submitted a retrospective analysis of accelerated hypofractionated Intensity modulated arc therapy (IMAT) using TomoTherapy in MPM following P/D or diagnostic biopsy. In the investigators experience of MPM, treatment of the intact lung with pleural IMAT using helical Tomotherapy is a safe and feasible option with an acceptable lung toxicity profile. The results obtained in terms of toxicity were encouraging. In fact, the investigators only observed one case of G3 pneumonia, and the patient in question is still alive and off oxygen therapy. Patient compliance with this short-course treatment was also very good.

Overall, the investigators found that accelerated hypofractionation with IMAT was feasible at the dose delivered and had an acceptable toxicity profile. So the investigators want to propose this protocol for treatment of MPM in intact lung to improve local control.

In patients with malignant pleural mesothelioma who underwent pleurectomy / decortications (P/D) or only diagnostic biopsy, it is difficult to deliver a tumoricidal dose of radiation to the pleura due to the presence of the ipsilateral lung. In recent years, the investigators have implemented a technique for irradiation of the pleura in intact lung, using accelerated hypofractionation with Tomotherapy in an attempt to reduce as far as possible, the dose to the ipsilateral lung. The aim of the treatment was palliation. The investigators analyzed the data of 36 patients with MPM, with a long follow-up without recording death cases related to radiation treatment or radiation pneumonitis grade 4.

In view of these data, the aim of this study is to increase the dose of treatment in patients suffering from MPM after P/D or biopsy.

The study will evaluate the feasibility of the treatment through the study of pulmonary acute and late toxicity; The treatment will be delivered using Tomotherapy that allows to adopt dose accelerated hypofraction criteria. Treatment duration is 5 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed MPM
2. Karnofsky Performance status scale 70-100 (see Appendix B)
3. Male or female, Aged >= 18 and ≤ 85 years
4. Life expectancy greater than 6 months
5. All clinical and pathological stage with the exclusion of contralateral mediastinum involvement (N3) and M1
6. Patients must have normal organ and marrow function as defined below:

   * leukocytes >3,000/microL
   * absolute neutrophil count >1,500/microL
   * platelets >100,000/microL
   * aspartate transaminase(AST)/alanine transaminase (ALT) <2.5 X institutional upper limit of normal
   * creatinine within normal institutional limits
   * glycemia < 100 mg/dl
7. Ability to understand and the willingness to sign a written informed consent document.
8. Forced expiratory volume in the 1st second(FEV1) ≥ 50
9. Patients after biopsy must have measurable disease defined as at least one lesion that can be accurately measured according to modified RECIST criteria; for resected patients no more than 3 months are allowed for RT start.
10. Written informed consent signed and dated before starting study procedure.
11. Female participants of child bearing potential and male participants whose partner is of child bearing potential must be willing to ensure that they or their partner use effective contraception during the study and for 4 months thereafter.

Exclusion Criteria:

1. Previous thorax radiotherapy
2. Chemotherapy is allowed but completed 3 weeks before RT starts
3. Participation in another clinical trial with any investigational agents within 30 days prior to study screening.
4. Patients with M1 have to be excluded to this study
5. FEV1 < 50
6. Age >85 years old
7. Respiratory needing oxygen therapy
8. Interstitial pneumopathy
9. Active pneumonitis
10. Fissural disease
11. Contralateral mediastinum involvement (N3) and M1
12. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | up to 36 months
  Acute and late toxicity evaluation by Common Terminology Criteria for Adverse Events (CTCAE) version 4.03, performing strumental tests (CT scan, spirometry) to evaluate adverse events including pulmonary toxicity

SECONDARY OUTCOMES:
Overall survival (OS) | up to 36 months
  time from randomization until death for any cause
Disease control rate (DCR) | up to 36 months
  the assessment of disease control rate (DCR) defined as proportion of patients with complete response (CR), partial response (PR) and stable disease (SD) for patients with evaluable disease using the Modified RECIST criteria for assessment of response in malignant pleural mesotelioma
time to progessione (TTP) | up to 36 months
  calculation of time to progression (TTP) for patients without evidence of disease or with not evaluable disease

CONTACTS AND LOCATIONS:
Overall Officials: Elisabetta Parisi, MD, Study Director — Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Via Maroncelli 40, 47014 Meldola, ITALY
Locations (1):
- SC Radiotherapy, Meldola, Italy

IPD SHARING:
Plan to Share IPD: Undecided